CLINICAL TRIAL: NCT01932697
Title: Phase II Evaluation of Adjuvant Hyperfractionated Radiation and Docetaxel for HPV Associated Oropharynx Cancer
Brief Title: Radiation Therapy and Docetaxel in Treating Patients With HPV-Related Oropharyngeal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1273; NCI-2013-01652 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1273 (Other: Mayo Clinic); 12-005272 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2013-08-27; First posted 2013-08-30 (Estimated); Results first posted 2019-09-18 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2023-09

CONDITIONS: Human Papillomavirus Infection; Stage I Oropharyngeal Squamous Cell Carcinoma; Stage II Oropharyngeal Squamous Cell Carcinoma; Stage III Oropharyngeal Squamous Cell Carcinoma; Stage IVA Oropharyngeal Squamous Cell Carcinoma; Stage IVB Oropharyngeal Squamous Cell Carcinoma
MeSH Terms: conditions — Papillomavirus Infections; Squamous Cell Carcinoma of Head and Neck | interventions — Docetaxel; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (docetaxel, hyperfractionated IMRT) (Experimental): Patients receive docetaxel IV over 1 hour on days 1 and 8 and undergo hyperfractionated IMRT BID 5 days a week on days 1-12 for a total of 20 fractions.
  Interventions: Drug: Docetaxel; Radiation: Hyperfractionation; Radiation: Intensity-Modulated Radiation Therapy; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment

INTERVENTIONS:
Drug: Docetaxel — Given IV
  Other Names: Docecad; RP56976; Taxotere; Taxotere Injection Concentrate
Radiation: Hyperfractionation — Undergo hyperfractionated IMRT
  Other Names: Hyperfractionated Radiation; Hyperfractionated Radiation Therapy; superfractionated radiation therapy
Radiation: Intensity-Modulated Radiation Therapy — Undergo hyperfractionated IMRT
  Other Names: IMRT; Intensity Modulated RT; Intensity-Modulated Radiotherapy
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This phase II trial studies how well radiation therapy and docetaxel work in treating patients with human papillomavirus (HPV)-related oropharyngeal cancer. Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving radiation therapy with docetaxel my kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the cumulative incidence of local/regional failure at 2 years after study registration.

SECONDARY OBJECTIVES:

I. To characterize the rate of acute grade 3 or higher functional mucosal adverse events (up to 1 month post-radiation therapy [XRT]) associated with adjuvant docetaxel + hyperfractionated radiotherapy (key secondary endpoint).

II. To assess changes in overall survival, disease-free survival, distant failure rates, and quality of life (QOL) associated with adjuvant docetaxel and hyperfractionated radiation.

III. To characterize other acute adverse events (up to 1 month post-XRT) and late grade 3 or higher non-hematologic adverse events (up to 2 years post-XRT) associated with adjuvant docetaxel + hyperfractionated radiotherapy.

TERTIARY OBJECTIVES:

I. To determine the genetic alterations of oropharynx tumor specimens and the detection rate of corresponding cell-free deoxyribonucleic acid (cfDNA) in the pre-surgical, post-surgical, and post-radiation blood of oropharynx cancer patients.

OUTLINE:

Patients receive docetaxel intravenously (IV) over 1 hour on days 1 and 8 and undergo hyperfractionated intensity-modulated radiation therapy (IMRT) twice daily (BID) 5 days a week on days 1-12 for a total of 20 fractions.

After completion of study treatment, patients are followed up at 14 days, 1 month, every 3 months for 2 years, every 6 months for 1 year and then annually for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* PRE-REGISTRATION
* Provide written informed consent
* Submission of research blood draw to be stored until after surgical resection of the primary tumor and confirmation of human papilloma virus (HPV) positivity (Mayo Clinic Rochester patients only)
* Patients with oropharynx carcinoma with a smoking history of ˂ 10 pack-year or equivalent 10 year history of tobacco product use and no recent history (within last 5 years) of tobacco use
* REGISTRATION
* Histological confirmation of HPV+ squamous cell carcinoma of the oropharynx; HPV positivity will be defined as positive staining for p16 on immunohistochemistry (IHC)
* Gross total surgical resection with curative intent of the primary tumor and at least unilateral neck dissection within 7 weeks of registration
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* Smoking history < 10 pack years or equivalent 10 year history of tobacco product use
* Absence of distant metastases on standard diagnostic work-up =< 10 weeks prior to registration; (chest computed tomography [CT], chest x-ray [CXR], positron emission tomography [PET]/CT, etc.)
* Must have one of the following risk factors:

  * Lymph node > 3 cm
  * 2 or more positive lymph nodes
  * Perineural invasion
  * Lymphovascular space invasion
  * T3 or microscopic T4a primary disease
  * Lymph node extracapsular extension
* Absolute neutrophil count (ANC) >= 1500/mm^3
* Platelet count >= 100,000/mm^3
* Hemoglobin >= 9.0 g/dL
* Direct bilirubin within upper limit of normal (ULN)
* Creatinine =< ULN x 1.5
* Negative pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Ability to complete questionnaire(s) by themselves or with assistance
* Provide informed written consent
* Willingness to return to enrolling institution for follow-up (during the active monitoring phase of the study)

Exclusion Criteria:

* Any significant tobacco history within the past five years
* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Immunocompromised patients and patients known to be human immunodeficiency virus (HIV) positive
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Other active malignancy =< 5 years prior to registration; EXCEPTIONS: non-melanotic skin cancer or carcinoma-in-situ of the cervix; NOTE: if there is a history or prior malignancy, they must not be receiving other specific treatment for their cancer
* History of myocardial infarction =< 180 days prior to registration, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* Prior history of radiation therapy to the affected site
* History of connective tissue disorders such as rheumatoid arthritis, lupus, or Sjogren's disease
* Presence of any of the following risk factors after surgery:

  * Any positive surgical margin
  * Adenopathy below the clavicles
* Prior systemic chemotherapy for the study cancer; NOTE: prior chemotherapy for a different cancer is allowable
* History of allergic reaction to docetaxel
* Receiving any medications or substances that are strong or moderate inhibitors of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4)

  * Use of strong or moderate inhibitors is prohibited =< 7 days prior to registration
* Receiving any medications or substances that are inducers of CYP3A4

  * Use of inducers is prohibited =< 12 days prior to registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2013-09-04 (Actual); Primary Completion 2016-10-20 (Actual); Study Completion 2021-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Ma, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic, Rochester, Minnesota

REFERENCES:
- [Derived] Ma DJ, Price KA, Moore EJ, Patel SH, Hinni ML, Garcia JJ, Graner DE, Foster NR, Ginos B, Neben-Wittich M, Garces YI, Chintakuntlawar AV, Price DL, Olsen KD, Van Abel KM, Kasperbauer JL, Janus JR, Waddle M, Miller R, Shiraishi S, Foote RL. Phase II Evaluation of Aggressive Dose De-Escalation for Adjuvant Chemoradiotherapy in Human Papillomavirus-Associated Oropharynx Squamous Cell Carcinoma. J Clin Oncol. 2019 Aug 1;37(22):1909-1918. doi: 10.1200/JCO.19.00463. Epub 2019 Jun 4. PMID 31163012

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A (Intermediate Risk): Patients received 30 Gy delivered in 1.5-Gy fractions twice per day over 2 weeks along with 15 mg/m2 docetaxel once per week.
- Cohort B (Extranodal Extension): Patients with extranodal extension who received the same treatment as Cohort A plus a simultaneous integrated boost to nodal levels with extranodal extension to 36 Gy in 1.8-Gy fractions twice per day.
Period: Overall Study
Arm/Group | Cohort A (Intermediate Risk) | Cohort B (Extranodal Extension)
Started | 38 | 43
Completed | 36 | 43
Not Completed | 2 | 0
Not completed — Received a different amount of tx | 1 | 0
Not completed — Ineligible | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A (Intermediate Risk) | Cohort B (Extranodal Extension) | Total
Number analyzed (Participants) | 36 | 43 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (6.7) | 58.9 (10.2) | 58.7 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 33 | 38 | 71
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 34 | 43 | 77
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group PS Scale: 0)Fully active, able to carry on all pre-disease performance without restriction; 1)Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2)Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours; 3)Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours; 4)Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair.
  Participants
    0 | 34 | 41 | 75
    1 | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: 2-year Loco-regional Tumor Control (LRC) Rate
Description: The 2-year loco-regional tumor control (LRC) rate (percentage) is defined as the percentage of patients with no local/regional recurrence or death 2 years after study registration.
Time Frame: 2 years
Measure: Number; unit: percentage of patients
Groups:
- Overall (Cohort A + Cohort B): Patients in Cohort A and Cohort B
Arm/Group | Cohort A (Intermediate Risk) | Cohort B (Extranodal Extension) | Overall (Cohort A + Cohort B)
Number analyzed (Participants) | 36 | 43 | 79
percentage of patients | 100 | 93 | 96.2

2. Secondary Outcome: Incidence of Grade 3 or Higher Mucositis Oral
Description: The overall percentage of patients experiencing grade 3 or higher mucositis oral graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 are reported below.
Time Frame: 4 months post-hyperfractionated radiation therapy
Measure: Number; unit: percentage of patients
Arm/Group | Cohort A (Intermediate Risk) | Cohort B (Extranodal Extension)
Number analyzed (Participants) | 36 | 43
percentage of patients | 8.3 | 4.7

3. Secondary Outcome: 2-year Overall Survival (OS) Rate
Description: The distribution of OS will be estimated using the method of Kaplan-Meier.
Time Frame: 2 years
Measure: Number; unit: percentage of patients
Groups:
- Cohort A: Patients received 30 Gy delivered in 1.5-Gy fractions twice per day over 2 weeks along with 15 mg/m2 docetaxel once per week.
- Cohort B: Patients with extranodal extension who received the same treatment as Cohort A plus a simultaneous integrated boost to nodal levels with extranodal extension to 36 Gy in 1.8-Gy fractions twice per day.
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 36 | 43
percentage of patients | 100 | 97.7

4. Secondary Outcome: 2-year Progression-free Survival (PFS)
Description: The distribution of PFS will be estimated using the method of Kaplan-Meier.
Time Frame: From registration to the first of either disease recurrence or death, assessed up to 2 years
Measure: Number; unit: percentage of patients
Arm/Group | Cohort A (Intermediate Risk) | Cohort B (Extranodal Extension)
Number analyzed (Participants) | 36 | 43
percentage of patients | 97.2 | 86.0

5. Secondary Outcome: 2-year Distant Metastasis-free Survival Rate
Description: The 2-year Distant metastasis-free survival rate (percentage) is defined as the percentage of patients with no distant recurrence or death 2 years after study registration.
Time Frame: 2 years
Measure: Number; unit: percentage of patients
Arm/Group | Cohort A (Intermediate Risk) | Cohort B (Extranodal Extension)
Number analyzed (Participants) | 36 | 43
percentage of patients | 97.2 | 88.4

6. Secondary Outcome: Change From Mean Baseline Score to Mean Score at 12 Months Post-RT in Swallow Function as Measured by the Pharyngeal Total Modified Barium Swallow Impairment Profile.
Description: The swallow evaluation consists of a modified barium swallow study(MBS), Functional Oral Intake Scale(FOIS), and Performance Status Scale Head & Neck(PSS-HN).The 17 swallow questions are rated using a 0 to 5 point scale, with 0 meaning no impairment and 5 max impairment. 6 questions produce a total oral score; scores from 10 questions produce a total pharyngeal score; 1 question produces an esophageal score.The PAS is a validated 8-point scale that ranks the depth of the bolus entry into the airway.A score of 1 indicates no airway entrance;score of 6+ indicate bolus passage past the vocal folds (aspiration).FOIS ranges from 1(nothing by mouth) to 7(total oral diet with no restrictions).PSS-H&N has 3 components:eating in public(0=always eat alone to 100=no restriction), understandability of speech(0=never understandable, score 100=always understandable), and normalcy of diet(score 0=tube fed to 100=full diet).These scores are summed and normalized to a 0 to 100 scale where 100 is best.
Time Frame: 12 months
Population: All patients that completed a Swallow Function assessment at baseline and 12-month post-RT were included. The difference in dose (30 vs 36 Gy) was not expected to have any appreciable difference in toxicity or PRO. What they represented were two different risk groups, hence the need to publish separate cohort disease control metric and why it makes less sense to sort out risk groups for radiation toxicity. It was pre-specified to report this analysis to compare timepoints and not cohorts.
Measure: Mean (Full Range); unit: score on a scale
Groups:
- All Patients: Cohort A and Cohort B were analyized together
Arm/Group | All Patients
Number analyzed (Participants) | 79
score on a scale
  Baseline time point | 5.57 [0 to 15]
  12 month time point | 4.48 [0 to 14]
Statistical Analysis 1: Comparison: All Patients; Test type: Superiority; p = .01, Paired t-test

7. Secondary Outcome: Functional Assessment of Cancer Therapy Head and Neck (FACT H& N) (Version 4)
Description: The FACT-H&N is a multidimensional, self-report QOL instrument specifically designed for use with head and neck cancer patients. It consists of 27 core items which assess patient function in four domains: Physical, Social/Family, Emotional, and Functional well-being, in addition to 12 site specific items to assess for head and neck related symptoms. Each item is rated on a 0 to 4 type scale where 4 is favorable and 0 unfavorable, and then combined to produce subscale scores for each domain, as well as a global QOL score- with possible score range from 0 to 156. Higher scores represent better QOL.
Time Frame: 1 year
Population: All patients treated per protocol and completed the FACT H&N forms were included in this analysis. The difference in dose (30 vs 36 Gy) was not expected to have any appreciable difference in toxicity or PRO. What they represented were two different risk groups, hence the need to publish separate cohort disease control metric and why it makes less sense to sort out risk groups for radiation toxicity. It was pre-specified to report this analysis to compare timepoints and not cohorts.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- All Patients: Both cohorts were combined for this analysis.
Arm/Group | All Patients
Number analyzed (Participants) | 68
score on a scale
  Baseline | 117.2 (17.7)
  12 months | 127.2 (17.7)
Statistical Analysis 1: Comparison: All Patients; Test type: Superiority; p < 0.001, Paired t-test

8. Secondary Outcome: European Organization for Research and Treatment for Cancer QOL Questionnaire for Head and Neck Cancer Module 35 (EORTC-QLQ HN35)
Description: QOL was measured by the European Organization for Research and Treatment for Cancer QOL Questionnaire for Head and Neck Cancer Module 35 (EORTC-QLQ HN35) at baseline and at 1-year post-treatment. Each question scores 0-4, with 0 being favorable and 4 being unfavorable. The average total score at baseline and average total score at 12 months post-RT is reported. The max total score possible is 140(Unfavorable) and the minimum total score possible is 0(Favorable). An increase in score indicates a greater quality of life A paired t-test compares the scores at these two timepoints.
Time Frame: 1 year post-treatment
Population: All patients treated per protocol and completed the EORTC-QLQ HN35 forms were included in this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort A (Intermediate Risk) | Cohort B (Extranodal Extension)
Number analyzed (Participants) | 36 | 43
score on a scale | 106.3 (10.7) | 111.4 (9.2)
Statistical Analysis 1: Comparison: Cohort A (Intermediate Risk) vs Cohort B (Extranodal Extension); Test type: Superiority; p < 0.001, Paired t-test

9. Secondary Outcome: EuroQol Five-dimensional Instrument (EQ-5D-3L)
Description: QOL was measured by the three-level version of the EuroQol five-dimensional instrument (EQ-5D-3L) at baseline and 1-year post-treatment. This consisted of 5 questions, each score 0 to 3 points with 3 being unfavorable and 0 being favorable. The total possible score per patient per time point is 15 and a minimum score of 0(favorable). The change in average total score at baseline and 12 months post-RT is reported. A paired t-test compares the scores at these two time points. A higher score indicates greater impairment.
Time Frame: 1 year post-treatment
Population: All patients who were treated per protocol and who completed a EQ-5D-3L were included in this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort A (Intermediate Risk) | Cohort B (Extranodal Extension)
Number analyzed (Participants) | 36 | 43
score on a scale | 6.3 (1.3) | 5.5 (0.9)
Statistical Analysis 1: Comparison: Cohort A (Intermediate Risk) vs Cohort B (Extranodal Extension); Test type: Superiority; p < 0.001, Paired t-test

10. Other Pre Specified Outcome: Changes in Transforming Growth Factor (TGF)-beta1 Levels
Description: These markers will be correlated with clinical endpoints like acute adverse events, cumulative incidence rates of local/regional failure, overall survival, and disease-free survival.
Time Frame: Baseline to 1 week post-radiation
Reporting Status: Not Posted

11. Other Pre Specified Outcome: E6/E7 Messenger Ribonucleic Acid (mRNA) of HPV16, Assessed on a Chromogenic RNA in Situ Hybridization (ISH) Assay Called RNAscope
Description: as for outcome 10
Time Frame: Baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 76 months
Description: All patients who received treatment and completed the adverse event form at least once are summarized below.
Arm/Group | Cohort A (Intermediate Risk) | Cohort B (Extranodal Extension)
All-Cause Mortality (participants affected / at risk) | 0/38 | 1/43
Serious Adverse Events (participants affected / at risk) | 5/38 | 5/43
Other Adverse Events (participants affected / at risk) | 38/38 | 43/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (Intermediate Risk) (N=38) | Cohort B (Extranodal Extension) (N=43)
Dysphagia (Gastrointestinal disorders) | 1 (2) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 2 (2) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bone infection (Infections and infestations) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (2)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Vasovagal reaction (Nervous system disorders) | 0 (0) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Lymphedema (Vascular disorders) | 2 (2) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (Intermediate Risk) (N=38) | Cohort B (Extranodal Extension) (N=43)
Dry mouth (Gastrointestinal disorders) | 37 (259) | 42 (305)
Dysphagia (Gastrointestinal disorders) | 28 (115) | 36 (130)
Esophagitis (Gastrointestinal disorders) | 14 (21) | 15 (25)
Mucositis oral (Gastrointestinal disorders) | 23 (35) | 28 (41)
Nausea (Gastrointestinal disorders) | 18 (25) | 13 (17)
Oral pain (Gastrointestinal disorders) | 20 (36) | 29 (56)
Fatigue (General disorders) | 34 (164) | 38 (139)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 3 (3) | 1 (2)
White blood cell decreased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Superficial soft tissue fibrosis (Musculoskeletal and connective tissue disorders) | 25 (115) | 31 (109)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (3) | 2 (7)
Stroke (Nervous system disorders) | 1 (1) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lymphedema (Vascular disorders) | 19 (76) | 26 (97)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-11-08): https://cdn.clinicaltrials.gov/large-docs/97/NCT01932697/Prot_SAP_000.pdf
  • Informed Consent Form (2017-06-05): https://cdn.clinicaltrials.gov/large-docs/97/NCT01932697/ICF_001.pdf